CLINICAL TRIAL: NCT00005451
Title: WINCATI Software Tool for Survey Research
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4384
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2000-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To design Computer Aided Telephone Interviewing (CATI) software tools for survey research.

DETAILED DESCRIPTION:
BACKGROUND:

CATI (Computer Aided Telephone Interviewing) became a primary means of obtaining quality epidemiological data. Its use steadily increased and in 1995 it was a major technology in use by almost every NIH Institute. Although CATI had been used for many years, its implementation had not kept up with technological developments in computers. Available CATI software products were deficient in features, inflexible, difficult to learn to use and had copious problems. Modern computer technology had the potential to satisfy the growing need for an improved product. This product had applications in over 3000 U.S. companies engaged in public opinion and market research.

DESIGN NARRATIVE:

In Phase I the investigators identified approaches that could be used to develop this software; justified and chose an approach; created requirements and designed specifications for the tool; developed a prototype; and produced a detailed project plan for implementation. In Phase II, the investigators completed and improved the prototype software and tested it in several areas

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-09; Study Completion 1999-07